CLINICAL TRIAL: NCT05202418
Title: Physiological Reactivity and Psychosocial Functioning in Pediatric Patients With Gastrointestinal Disease
Brief Title: Stress in Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Bonney Reed, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00085974; 5K23DK122115-02 (NIH); 1R03DK136975-01 (NIH)
Record Dates: First submitted 2021-12-09; First posted 2022-01-21 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases; Psychological
Keywords: skin conductance reactivity; Systemic inflammation
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback Enhanced Treatment (Experimental): Participants in this group will participate in biofeedback enhanced cognitive behaviorally based coping skills treatment. Treatment will consist of a 6-visit group intervention conducted online, via Emory zoom. Groups will include 5-8 patients each. Sessions will include brief, daily homework to facilitate mastery that is developmentally tailored to youth (e.g., practice skills with support from phone or tablet apps). Groups will meet approximately every week for 6 weeks. Advanced Ph.D. students in clinical psychology and Principal Investigator will deliver the treatment protocol. They will complete questionnaires before and after each session to measure autonomic reactivity in response to stress induction and coping strategies.
  Interventions: Behavioral: Biofeedback Enhanced Treatment
- Wait-list control (No Intervention): Participants randomized to the wait-list control group will complete the same measures of lifetime stress, autonomic reactivity, depression, anxiety. The identical treatment will be offered to control participants after the 6-week time point.

INTERVENTIONS:
Behavioral: Biofeedback Enhanced Treatment — The intervention involves biofeedback enhanced cognitive behaviorally based coping skills treatment. Treatment will consist of a 6-visit group intervention conducted online, via Emory zoom. Groups will include 5-8 patients each. Sessions will include brief, daily homework to facilitate mastery that is developmentally tailored to youth (e.g., practice skills with support from phone or tablet apps). Groups will meet approximately every week for 6 weeks. Advanced Ph.D. students in clinical psychology and Principal Investigator will deliver the treatment protocol. Participants will complete questionnaires before and after each session to measure autonomic reactivity, lifetime stress, depression, anxiety in response to stress induction, and coping strategies.
  Other Names: Behavioral Intervention
  Arms: Biofeedback Enhanced Treatment

SUMMARY:
This is a prospective, assessment-based study to examine the relationship between psychophysiological functioning and psychological symptoms in youth newly diagnosed with inflammatory bowel disease (IBD) compared to healthy controls.

DETAILED DESCRIPTION:
Similar to other chronic stressors, diagnosis with a chronic illness places youth at risk of adverse psychosocial outcomes. Inflammatory bowel diseases (IBD), Crohn's disease, ulcerative colitis, and indeterminate colitis are chronic, immune-mediated diseases of the gastrointestinal tract characterized by unpredictable remissions of disease activity followed by relapses of symptoms. Although some research has found higher levels of disease activity to relate to greater depressive symptoms, the overall relationship between disease activity and emotional functioning has been mixed, suggesting that additional individual differences need to be considered in addition to illness-related factors when predicting emotional outcomes. Increased risk for developing anxiety disorders and depression has been documented in youth with IBD. Individual differences in physiological reactivity may affect patients' risk for developing psychosocial difficulties within the context of chronic stress. Additional risk factors for developing psychosocial challenges need to be identified to identify moderators of outcomes above and beyond disease activity.

Individual differences in physiological reactivity may affect patients' risk for developing psychosocial difficulties within the context of chronic stress. Physiological reactivity, which broadly refers to bodily reactions in response to a stressor, varies with regards to intensity and threshold for activation between individuals.

In youth affected by non-medical chronic stress (e.g., family conflict, trauma history), measures of autonomic dysfunction have been used to explain why some individuals have worse psychological and physical outcomes compared to others exposed to similar levels of chronic stress. Results support autonomic dysfunction as a vulnerability factor for adjustment problems within the context of chronic environmental stress.

The current study aims to test whether differences in psychophysiological reactivity serve as risk factors in the relationship between clinical disease activity in youth newly diagnosed with IBD and psychosocial adjustment problems. The relationship between psychophysiological reactivity and psychosocial adjustment problems in youth with IBD will be compared to healthy controls. Youth participants with IBD will be enrolled in a coping skills treatment to test the effectiveness of a cognitive-behavioral intervention including biofeedback to reduce anxiety and depression and disease symptoms. The research team will conduct a pilot intervention targeting autonomic dysfunction through biofeedback-enhanced coping skills treatment delivered virtually over 6-sessions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with biopsy-confirmed IBD
* Ages 13 through 18 years inclusive
* English fluency for parent and child participants.
* Accompanied by at least 1 parent/guardian who is willing to participate
* Positive depression or anxiety symptom screen using the patient health questionnaire (PHQ-9) or Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Anxiety measures

Exclusion Criteria:

* Previous diagnosis of intellectual disability
* Autism spectrum disorder.
* Parent is unwilling to participate.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2024-01-13 (Actual); Study Completion 2024-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Reed, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Atlanta Metropolitan Area, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory Children's Center Building, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The research team will share individual participant data that underlie the results reported in a published article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: The research team will share the data beginning 6 months and ending 36 months following article publication.
Access Criteria: The research team will share the data with researchers, who provide a methodologically sound proposal. Data will be shared to achieve aims in the approved proposal All requests and proposals should be directed to ebreed@emory.edu up to 36 months following article publication.

REFERENCES:
- [Derived] Younginer ST, Westbrook A, Buzenski J, Dykes C, Kugathasan S, Talmadge C, Reed B. Health-related quality of life in youth with chronic gastrointestinal disease following a biofeedback enhanced cognitive behavioral therapy intervention: A randomized controlled trial. J Pediatr Gastroenterol Nutr. 2026 Jan 4. doi: 10.1002/jpn3.70333. Online ahead of print. PMID 41486461

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Children's Healthcare of Atlanta (CHOA) at Egleston in Atlanta, Georgia, USA. Participant enrollment began on February 27, 2022, and 3 rounds of treatment and paired waitlist groups were held. All follow-ups were complete by January 13, 2024.
Pre-assignment Details: Participants in the waitlist control group completed lifetime stress, autonomic reactivity, depression, and anxiety surveys at baseline and 6 weeks. A 2-month follow-up was not conducted during the waitlist period, as the biofeedback intervention was given after 6 weeks. After completing the Biofeedback Enhanced Treatment, participants took part in the 2-month follow-up assessments. All 2-month follow-up data were then combined and analyzed for both groups.
Groups:
- Biofeedback Enhanced Treatment: Participants will engage in biofeedback-enhanced, cognitive-behavioral coping skills treatment. Sessions will include brief, daily homework assignments tailored to youth (e.g., using apps for skill practice). Participants will complete pre- and post-session questionnaires to assess autonomic reactivity, lifetime stress, depression, anxiety, and coping strategies in response to stress induction.
  Biofeedback Enhanced Treatment: The intervention involves biofeedback enhanced cognitive behaviorally based coping skills treatment. Treatment will consist of a 6-visit group intervention conducted online, via Emory Zoom. Groups will include 5-8 patients each. Sessions will include brief, daily homework to facilitate mastery, developmentally tailored to youth (e.g., practice skills with support from phone or tablet apps). Groups will meet approximately every week for 6 weeks. Advanced Ph.D. students in clinical psychology and the Principal Investigator will deliver the treatment protocol. Participants will complete questionnaires before and after each session to measure autonomic reactivity, lifetime stress, depression, anxiety in response to stress induction, and coping strategies.
- Wait-list Control: Participants randomized to the wait-list control group will complete the same measures of lifetime stress, autonomic reactivity, depression, and anxiety. The intervention was offered to control participants after the 6-week time point, and all 2-month follow-up surveys and assessments were completed only after finishing the Biofeedback Enhanced Treatment.
Period: Overall Study
Arm/Group | Biofeedback Enhanced Treatment | Wait-list Control
Started | 26 (For participants randomized to the treatment group, clinical assessments, including study questionnaires and the HRV assessment, were conducted at baseline (within 1 week before starting treatment), at the end of treatment (6 weeks after baseline), and all other assessments were completed 14 weeks after baseline to capture the 2-month follow-up after treatment.) | 27 (Participants randomized to the waitlist control group completed the same assessment protocol at the time of randomization (Baseline) and again 6 weeks later.)
Completed | 23 | 25 (The biofeedback enhancement intervention was administered after 6 weeks. After completing the Biofeedback Enhanced Treatment, participants completed satisfaction and HRV assessments at the 6-week and 2-month follow-up points, after finishing the treatment.)
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofeedback Enhanced Treatment | Wait-list Control | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.58 (1.38) | 15.37 (1.45) | 15.00 (1.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 7 | 13 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 24 | 26 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 23 | 22 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 27 | 51
Inflammatory Bowel Disease (IBD) Diagnosis [Count of Participants; unit: Participants]
  Crohn's Disease | 16 | 20 | 36
  Ulcerative Colitis | 8 | 6 | 14
  Indeterminate Colitis | 0 | 1 | 1
Time since diagnosis [Mean (Standard Deviation); unit: years] | 2.88 (2.57) | 3.53 (2.80) | 3.22 (2.69)
Estimated household yearly income before taxes [Count of Participants; unit: Participants]
  $25,000 to $49,999 | 2 | 0 | 2
  $50,000 to $74,999 | 3 | 1 | 4
  $75,000 to $99,999 | 2 | 5 | 7
  $100,000 to $124,999 | 6 | 4 | 10
  $125,000 to $149,999 | 1 | 4 | 5
  Above $150,000 | 10 | 11 | 21
  Not Reported | 1 | 1 | 2
Caregiver relationship to the child [Count of Participants; unit: Participants]
  Mother | 24 | 22 | 46
  Father | 0 | 3 | 3
  Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Retention Rate
Description: Retention rates will be summarized using the number of individuals who gave consent to participate in the trial, who completed 6 weeks of the intervention they were randomized to, as well as the count of participants completing the Post-Treatment assessment 2 months after finishing 6 weeks of Biofeedback Enhanced Treatment.
Time Frame: 6 weeks (End of treatment), and 2 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Biofeedback Enhanced Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 27
Participants
  Retention at 6 weeks (End of treatment) | 23 | 25
  Retention at 2 months post-treatment | 19 | 22

2. Primary Outcome: Client Satisfaction Questionnaire (CSQ-8) Scores Following Biofeedback Enhanced Treatment
Description: Acceptability of the Biofeedback Enhanced Treatment was assessed using adolescent- and parent-reported program satisfaction ratings on the Client Satisfaction Questionnaire (CSQ-8). Adolescents and parents completed this 8-item survey on a 4-point scale, with total scores ranging from 8 to 32; higher scores indicated greater satisfaction. Each group completed the questionnaire 6 weeks after finishing the Biofeedback Enhanced Treatment. No survey was provided to participants during the waitlist phase, as no treatment was administered during the waiting period.
Time Frame: 6 weeks (End of treatment)
Population: Satisfaction data applies only to the Biofeedback Enhanced Treatment (BET), as the control group did not receive treatment during the first 6 weeks. Satisfaction was assessed after both groups had completed their treatments, and the data were combined for analysis. These results include data from participants who completed the Biofeedback Enhanced Treatment and the satisfaction surveys 6 weeks post-treatment (BET), with data from both groups analyzed after treatment completion.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Biofeedback Enhanced Treatment and Waitlist Control After Completing Treatment: All participants randomized to either the Biofeedback Enhanced Treatment group or the Waitlist Control group were evaluated and analyzed together after completing treatment within their respective periods.
Arm/Group | Biofeedback Enhanced Treatment and Waitlist Control After Completing Treatment
Number analyzed (Participants) | 42
score on a scale
  Child Report at 6 weeks (End of treatment) | 28.02 (2.90)
  Parent Report at 6 weeks (End of treatment) | 28.73 (3.18)

3. Secondary Outcome: Change in the Children's Depression Inventory 2 (CDI-2) at Six Weeks Compared to Baseline
Description: Children's Depression Inventory 2 (CDI-2) is a child-report measure of physiological, behavioral, and emotional symptoms of depression. It is a widely used tool for assessing depressive symptoms in children and adolescents. It includes 28 items, each with three possible responses that reflect different levels of severity: 0 (absence of symptoms), 1 (mild or probable symptom), or 2 (definite symptom). Raw scores are converted to t-scores ranging from 0 to 100, with a mean of 50 and a standard deviation of 10. A decrease in the score indicates an improvement in depressive symptoms (depressive symptoms decrease over time).
Time Frame: 6 weeks (End of treatment)
Population: This analysis includes participants who completed the baseline survey.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Biofeedback Enhanced Treatment | Wait-list Control
Number analyzed (Participants) | 24 | 27
T-score | -1.99 [-4.49 to 0.47] | 0.00 [-2.18 to 2.18]

4. Secondary Outcome: Change in the Children's Depression Inventory 2 (CDI-2) at 2 Months Post-treatment Compared to Baseline
Description: Children's Depression Inventory 2 (CDI-2). The CDI 2 is a child-report measure of physiological, behavioral, and emotional symptoms of depression. The full-length CDI 2: Self-Report (CDI 2:SR) is a 28-item assessment that yields a Total Score, two scale scores, and four subscale scores. For each item, the respondent is presented with three choices that correspond to three levels of symptomatology: 0 (absence of symptoms), 1 (mild or probable symptom), or 2 (definite symptom). Raw scores are converted to t-scores ranging from 0 to 100, with a mean of 50 and a standard deviation of 10. A decrease in the score indicates an improvement in depressive symptoms (depressive symptoms decrease over time).
Time Frame: 2 months post-Biofeedback Enhanced Treatment
Population: The results include data from participants in both groups after completing the Biofeedback Enhanced Treatment. No 2-month follow-up data were collected from the control group during the waiting period, as they received the intervention at 6 weeks. Data were collected 2 months after completing the treatment in each group, and these were combined for analysis, as specified in the protocol, which outlines that the changes will be summarized within groups.
Measure: Mean (95% Confidence Interval); unit: T-score
Groups:
- Biofeedback Enhanced Treatment and Waitlist Control After Completing Treatment: All participants randomized to either the Biofeedback Enhanced Treatment group or the Waitlist Control group were evaluated and analyzed together after completing the treatment within their respective periods. Both groups were combined for analysis at the 2-month follow-up after each group completed the Biofeedback Enhanced Treatment in different periods.
Arm/Group | Biofeedback Enhanced Treatment and Waitlist Control After Completing Treatment
Number analyzed (Participants) | 51
T-score | -4.17 [-6.63 to -1.71]

5. Secondary Outcome: Changes in the Behavior Assessment System for Children (BASC) Depression Parent Rating Scale at 6 Weeks
Description: Depressive symptoms were assessed using the 13-item Depression subscale of the Behavior Assessment System for Children, 3rd Edition (BASC-3). The BASC-3 Parent Rating Scale (PRS) is a tool used to evaluate problem behaviors, including internalizing, externalizing, and adaptive behaviors. Parents rate the frequency of these behaviors on a scale from 'Never' to 'Almost Always.' T-scores are used to compare responses to normative data for children of the same age and gender. Raw scores are converted to t-scores ranging from 0 to 100, with a mean of 50 and a standard deviation of 10. A decrease in the score indicates an improvement in depressive symptoms (depressive symptoms decrease over time).
Time Frame: baseline, 6 weeks (End of treatment)
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Biofeedback Enhanced Treatment | Wait-list Control
Number analyzed (Participants) | 24 | 27
T-score | -3.64 [-7.21 to -0.07] | 0.44 [-2.88 to 3.76]

6. Secondary Outcome: Changes in the Behavior Assessment System for Children (BASC) Depression Parent Rating Scale at 2 Months After Completing Treatment Intervention
Description: as for outcome 5
Time Frame: baseline, 2 months post-treatment
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Biofeedback Enhanced Treatment and Waitlist Control After Completing Treatment
Number analyzed (Participants) | 51
T-score | -4.60 [-7.06 to -2.15]

7. Secondary Outcome: Changes in the Screen for Child Anxiety Related Disorders (SCARED) Scores at 6 Weeks (End of Treatment)
Description: The Screen for Child Anxiety Related Disorders (SCARED) is a 41-item inventory rated on a 3-point Likert scale (0 "Not true or hardly ever true" to 2 "Very true or often true") used to screen for anxiety disorders. It provides a Total score and scores across five domains: panic/somatic, separation anxiety, generalized anxiety, social anxiety, and school phobia. The total score ranges from 0 to 82, with higher scores indicating greater anxiety. A score of 25 or higher may suggest an anxiety disorder, while scores above 30 are more specific. A decrease in score reflects symptom improvement.
Time Frame: baseline, 6 weeks (End of treatment)
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Biofeedback Enhanced Treatment | Wait-list Control
Number analyzed (Participants) | 24 | 27
Score on a scale
  Child Report at 6 weeks (End of treatment) | -5.05 [-9.69 to -.04] | -0.67 [-4.8 to 3.47]
  Parent Report 6 weeks (End of treatment) | -1.87 [-5.87 to 2.13] | -1.84 [-5.53 to 1.85]

8. Secondary Outcome: Changes in Screen for Child Anxiety Related Disorders (SCARED) Scores in Both Groups at 2 Months After Completing Treatment
Description: as for outcome 7
Time Frame: baseline, 2 months post treatment
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Biofeedback Enhanced Treatment and Waitlist Control After Completing Treatment
Number analyzed (Participants) | 51
Score on a scale
  Child Report at 2 months post treatment (End of treatment) | -4.28 [-7.14 to -1.42]
  Parent Report at 2 months post treatment | -1.87 [-5.87 to 2.13]

9. Secondary Outcome: Changes in the Children's Somatic Symptoms Inventory (CSSI) 7-item (GI Subscale) After Completion of Biofeedback Enhanced Treatment
Description: Self-report of disease activity using the Children's Somatic Symptoms Inventory (CSSI) 7-item (GI Subscale), will be collected. The GI symptom subscale includes items on nausea, constipation, diarrhea, abdominal pain, vomiting, bloating, and food-induced discomfort. Each item asks the child to rate the frequency and intensity of symptoms over a specific period (e.g., "In the past week, how often have you felt stomachaches?"). Response options include: 0 - "Not at all"; 1 - "A little bit"; 2 - "Somewhat"; 3 - "Quite a bit"; 4 - "Very much." Scores are summed to obtain a total score for gastrointestinal symptoms. High scores, indicating frequent or intense gastrointestinal complaints, may suggest significant distress or a need for intervention. A decrease in the score reflects symptom improvement.
Time Frame: baseline, 6 weeks (End of treatment)
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Biofeedback Enhanced Treatment | Wait-list Control
Number analyzed (Participants) | 24 | 27
Score on a scale
  Child Report at 6 weeks (End of treatment) | -1.29 [-2.91 to 0.32] | 0.56 [-0.88 to 1.99]
  Parent Report at 6 weeks (End of treatment) | -2.79 [-4.53 to -1.04] | -0.12 [-1.73 to 1.49]

10. Secondary Outcome: Changes in the Children's Somatic Symptoms Inventory- (CSSI) 7-item (GI Subscale) at 2 Months After Completion of Treatment Intervention
Description: Self-report of disease activity using the Children's Somatic Symptoms Inventory-(CSSI) 7-item (GI Subscale) will be collected from parents and teens. The GI symptom subscale includes items on nausea, constipation, diarrhea, abdominal pain, vomiting, bloating, and food-induced discomfort. Each item asks the child to rate the frequency and intensity of symptoms over a specific period (e.g., "In the past week, how often have you felt stomachaches?"). Response options include: 0 - "Not at all"; 1 - "A little bit"; 2 - "Somewhat"; 3 - "Quite a bit"; 4 - "Very much." Scores are summed to get a total gastrointestinal score. High scores, indicating frequent or intense symptoms, may suggest significant distress or the need for intervention. A decrease in score reflects symptom improvement.
Time Frame: baseline, 2 months post-treatment
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Biofeedback Enhanced Treatment and Waitlist Control After Completing Treatment Intervention: All participants randomized to either the Biofeedback Enhanced Treatment group or the Waitlist Control group were evaluated and analyzed together after completing the treatment within their respective periods. Both groups were combined for analysis at the 2-month follow-up after each group completed the Biofeedback Enhanced Treatment in different periods.
Arm/Group | Biofeedback Enhanced Treatment and Waitlist Control After Completing Treatment Intervention
Number analyzed (Participants) | 51
Score on a scale
  Child Report at 2 months post-treatment(End of treatment) | 0.62 [-0.69 to 1.94]
  Parent Report at 2 months post-treatment (End of treatment) | -0.01 [-1.27 to 1.25]

11. Secondary Outcome: Change in Autonomic Reactivity at 6 Weeks (End of Treatment)
Description: Autonomic reactivity will be measured using Heart Rate Variability (HRV) with the Inner Balance system by HeartMath. HRV will be assessed before treatment, post-treatment, and at follow-up. The mediation effect will be estimated using the difference in regression coefficients (β1 - β2). Adolescent HRV data was collected via the InnerBalance sensor during the pre-treatment (T1) and post-treatment (T2) assessments.
  The RR interval represents the time between heartbeats, while the NN interval normalizes this time, accounting for noise or artifacts. HRV measures, including the standard deviation of NN intervals (SDNN) and the root mean square of successive RR interval differences (RMSSD), are calculated from these intervals. Higher values of SDNN and RMSSD are considered more adaptive.
Time Frame: baseline, 6 weeks (End of treatment)
Measure: Mean (95% Confidence Interval); unit: milliseconds (ms)
Arm/Group | Biofeedback Enhanced Treatment | Wait-list Control
Number analyzed (Participants) | 24 | 27
milliseconds (ms)
  SDNN at 6 weeks (End of treatment) | 15.6 [-2.12 to 33.32] | 16.74 [0.99 to 32.49]
  RMSSD at 6 weeks (End of treatment) | -4.09 [-27.64 to 19.47] | 16.02 [-4.86 to 36.91]

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from the time consent was given to participate in the study through 2 months post-treatment.
Arm/Group | Biofeedback Enhanced Treatment | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 0/24 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT05202418/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT05202418/ICF_000.pdf